CLINICAL TRIAL: NCT00482651
Title: Imaging of Vulnerable Plaques in Coronary Artery Disease by Multidetector Computed Tomography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Danish Research Agency (Other); Philips Medical Systems (Industry); Danish Heart Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MDCT2403
Record Dates: First submitted 2007-06-04; First posted 2007-06-05 (Estimated); Last update posted 2012-01-23 (Estimated); Status verified 2012-01

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis | interventions — Ultrasonography, Interventional; Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- UAP, SAP (Experimental)
  Interventions: Radiation: Multidetector computed tomography scanning; Procedure: Coronary angiography (CAG); Procedure: Intravascular ultrasound; Procedure: Blood sample

INTERVENTIONS:
Radiation: Multidetector computed tomography scanning — contrast Multidetector CT-scanning
  Other Names: Philips Brilliance 64
Procedure: Coronary angiography (CAG) — CAG and if necessary PCI. Included patients are already assigned for CAG
Procedure: Intravascular ultrasound — During CAG Intravascular Ultrasound will be performed in the three coronary arteries
  Other Names: Volcano / virtual histology
Procedure: Blood sample — a blood sample at baseline after 3 months and at the end of the follow up (after 12 months)

SUMMARY:
Atherosclerosis is a chronic and multifocal immunoinflammatory, fibroproliferative disease of medium-sized and large arteries driven by lipid. Atherosclerosis is rarely fatal unless thrombosis supervene, causing an acute coronary syndrome. Therefore, for event-free survival, the vital question is not why atherosclerosis develops but rather why atherosclerosis, after years after indolent growth, suddenly becomes complicated with luminal thrombosis.

The great majority of coronary plaques will remain quiescent, at least from a clinical point of view.

Acute coronary syndrome is primarily precipitated by a ruptured plaque. The precipitating factor or condition may be found outside rather than inside the plaque.

The challenge is to find the plaque(s) destined for the next thrombus-mediated heart attack(s), treat, and thus avoid the heart attack(s). Identification of vulnerable plaques has become a key issue. The natural history of individual plaques (risk of thrombosis) is unknown and needs to be established.

Multidetector computed tomography (MDCT) can provide angiography and imaging of the vessel wall (detection, quantification and characterization of plaques).

The intention of this project is to evaluate the accuracy of coronary MDCT in identifying and differentiating the morphology of coronary atherosclerotic plaques.

DETAILED DESCRIPTION:
Atherosclerosis without thrombosis is rarely fatal. It is the acute thrombotic complications which account for disability and death. Therefore, for event-free survival, the question is not why atherosclerosis develops but rather why atherosclerosis, after years after indolent growth, suddenly becomes complicated with luminal thrombosis.

Post-mortem and clinical observations indicate that patients with acute coronary syndromes often have many ruptured and/or active plaques in their coronary arteries.

The challenge is to find the plaque(s) destined for the next thrombus-mediated heart attack(s), treat, and thus avoid the heart attack(s). Identification of vulnerable plaques have become a key issue. The natural history of individual plaques (risk of thrombosis) is unknown and needs to be established. Multidetector computed tomography (MDCT) can provide angiography and imaging of the vessel wall.

Hypothesis:

It is by CT-scanning possible to 1a) identify and differentiate the morphology of coronary atherosclerotic plaques.

1b) identify vulnerable plaques.

Materials and methods:

1. Development of an MDCT scan protocol for accurate assessment of coronary artery plaque composition by ex vivo examination of human coronary arteries from the Institute of Forensic Medicine, University of Aarhus. Scan protocols parameters and intravascular contrast material will be varied to optimize accurate assessment of coronary plaque composition. MDCT will be compared to histopathology.
2. A cross-sectional study with clinical application of the efficiency parameters defined in sub-study 1. Forty consecutive patients with non ST-elevation myocardial infarction/unstable angina, and 80 consecutive patients with stable angina will be recruited and investigated with MDCT followed by CAG with IVUS/virtual histology.
3. A prospective, longitudinal study. After a period of 12 months all patients from sub-study 2 will be re-investigated.
4. Before the cross-sectional study a small pilot-study will be performed. Ten patients with non ST-elevation myocardial infarction/unstable angina will undergo MDCT and CAG with IVUS/virtual histology. These patients will after one months undergo another MDCT. This is done to make sure that it is possible to perform the planned longitudinal study.

Research plan:

1. Development of an MDCT scan protocol for accurate assessment of coronary artery plaque composition.
2. Clinical application of the MDCT scan protocol for in vivo differentiation of coronary artery plaque morphology. Morphologic findings will be categorized and compared with IVUS/virtual histology for confirmation.
3. Re-evaluation of plaque density and morphology one year after inclusion by a second in vivo contrast-enhanced MDCT-scanning to define which morphological plaque categories are at risk of progression.

ELIGIBILITY:
Inclusion Criteria:

* Unstable angina pectoris Stable angina pectoris

Exclusion Criteria:

* known allergy towards the contrast agent not able to hold ones breath for 20 seconds pulmonal, renal or heart failure, cancer, or inflammatory disease arrythmia intolerant to treatment with beta-blockers claustrophobia, pregnancy, breast-feeding previous bypass surgery or PCI continuing breast pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2007-11; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Ability to identify and characterise atherosclerotic plaques by multidetector CT | immediately after the CT-scanning

SECONDARY OUTCOMES:
The impact of different CT-parameters on the ability to identify and characterise atherosclerotic plaques | immediately after the CT-scanning
the growth/development of atherosclerosis | one year

CONTACTS AND LOCATIONS:
Overall Officials: Hans Erik Boetker, MD,PhD,DMSc, Study Director — Aarhus University Hospital
Locations (1):
- Department of Cardiology, Aarhus University hospital, Skejby, Aarhus N, Denmark